CLINICAL TRIAL: NCT05612893
Title: Discover the Immune Signature of Sepsis Caused by Acute Pulmonary Infection: A Cohort Study
Acronym: DISPLAY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Bin Cao, Professor, Capital Medical University
Other Study IDs: 2021-I2M-1-048
Record Dates: First submitted 2022-11-02; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Sepsis; Viral Pneumonia; Influenza; Upper Respiratory Tract Infection
MeSH Terms: conditions — Sepsis; Pneumonia, Viral; Influenza, Human; Respiratory Tract Infections | interventions — Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood was collected by the hospital nurse. Nasal mucosal cells will be obtained by Nasal Cytology Curettes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Influenza upper respiratory infection: This cohort aims to descirbe the nasal mucosal immune response in influenza patients. We will collect nasal mucosal cells from influenza patients using Nasal Cytology Curettes. Blood samples will also be obtained from the patient. All samples will be used for single cell sequencing.
  Interventions: Other: pathogen
- Viral Sepsis and Viral pneumonia: The purpose of this cohort is to characterize the immune pattern of patients with viral sepsis and find specific target for the treatment of viral sepsis. Blood samples will be obtained from the viral sepsis/pneumonia patients.All samples will be used for transcriptome sequencing.
  Interventions: Other: pathogen
- Bacterial Sepsis and Bacterial pneumonia: This cohort served as a control for the viral sepsis/pneumonia cohort.Blood samples will be obtained from the bacterial sepsis/pneumonia patients.All samples will be used for transcriptome sequencing.
  Interventions: Other: pathogen

INTERVENTIONS:
Other: pathogen — The patients were divided into groups according to the pathogen(bacteria or virus).
  The influenza upper respiratory tract infection cohort will be grouped mainly according to age.
  Other Names: age

SUMMARY:
The goal of this observational study is to describe the immune signature of acute pulmonary infection.The main questions it aims to answer are:

1. Nasal mucosal immune response in patients with influenza infection
2. Difference of immune response between Viral sepsis and Bacterial sepsis
3. Immunological differences between Viral sepsis and Viral pneumonia

DETAILED DESCRIPTION:
1. Aging could influence host immune response. Elderly people are more likely to progress to severe pneumonia than young people. Nasal mucosa is the initial infection site of influenza infection. Single cell sequencing of nasal mucosal cell that may provide valuable insights into host response to influenza infection.
2. Sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection. Although bacteria are considered as the main pathgens of sepsis，SARS-CoV-2 or influenza infection also can cause multiple organ dysfunction which meet the definition of Sepsis 3.0. Viral sepsis has not received enough attention for a long time. It is important to understand the difference between viral sepsis and bacterial sepsis that may help to develop better strategies to diagnose and treat sepsis.
3. Viral pneumonia is one of the leading infectious cause of death woldwide.Pneumina is the most common cause of sepsis.The mechanism of viral pneumonia progressing to sepsis needs to be further investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at time of signing Informed Consent Form
2. chest imaging confirmed pneumonia.
3. Informed consent is obtained
4. The pneumonia onset ≤8 days

Exclusion Criteria:

1. SaO2/SPO2≤94% on room air or Pa02/Fi02 ratio <300mgHg before the onset of pneumonia
2. Severe liver disease (e.g. Child Pugh score ≥ C, AST>5 times upper limit)
3. Patients with known severe renal impairment (estimated glomerular filtration rate ≤30 mL/min/1.73 m2) or receiving continuous renal replacement therapy, hemodialysis,peritoneal dialysis）
4. Pregnant Or Lactating Women
5. Patients were eligible for organ transplantation or had undergone previous organ transplantation surgery
6. HIV infection
7. Had unstable angina or myocardial infarction within 30 days without vascular recanalization treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed pneumonia and signed informed consent will be enrolled.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-16 (Estimated); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
upper respiratory infection or pneumonia or Sepsis | up to 28 days
  Patients were grouped and compared according to their diagnosis.

SECONDARY OUTCOMES:
Clinical status | days 0, 3, 7
  assessed by Sequential Organ Failure Assessment
All cause mortality | up to 28 days
Length of hospital stay (days) | up to 28 days
Length of ICU stay (days) | up to 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We will share the transcriptome data with other researchers.
Supporting Information: Study Protocol, ICF, Analytic Code